CLINICAL TRIAL: NCT07269171
Title: Evaluation of the Effects of Dietary Supplements Containing Trypsin, Chymotrypsin and Serratia Peptidase on Postoperative Edema, Pain and Trismus After Mandibular Impacted Third Molar Extraction.
Brief Title: The Effect of Supplementary Foods Containing Trypsin, Chymotrypsin and Serratia Peptidase on Healing After Impacted Wisdom Tooth Surgery
Acronym: Trypsin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özgün Yıldırım, Doctor, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15.05.2025-2025/9-9/11
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Oral Health Care
Keywords: nutritional supplements; oral and maxillofacial surgery; wisdom teeth; trypsin, chymotrypsin and serratia peptidase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients undergoing right mandibular third molar surgery will receive standard postoperative medication: painkillers (dexketoprofen 25 mg), antibiotics (amoxicillin 875 mg + clavulanic acid 125 mg), and a chlorhexidine 0.12% + benzydamine 0.15% mouthwash. Demographic data will be recorded preoperatively. All surgeries will be performed under sterile conditions with inferior alveolar nerve block and buccal infiltration using articaine 4% with epinephrine 1:100,000. Operation time will be measured from incision to last suture. Osteotomy and, when necessary, tooth sectioning will be performed with a surgical handpiece and saline irrigation. After extraction, sockets will be smoothed and closed with 3-0 silk sutures. Patients will be reviewed on postoperative days 1, 2, 3, and 7, and pain, edema, and trismus will be recorded.
  Interventions: Procedure: Pain Assessment; Procedure: Number of Analgesics Needed; Procedure: Edema Assessment; Procedure: Trismus Assessment
- Control group (Experimental): Patients undergoing right mandibular third molar surgery will receive standard postoperative medication, including dexketoprofen 25 mg, amoxicillin 875 mg + clavulanic acid 125 mg, and a 0.12% chlorhexidine + 0.15% benzydamine mouthwash. Demographic data will be recorded preoperatively. All operations will be performed under sterile conditions with inferior alveolar nerve block and buccal infiltration using 4% articaine with 1:100,000 epinephrine. Surgical time will be measured from incision to final suture. Osteotomy and, when required, tooth sectioning will be performed with a surgical handpiece and saline irrigation. After extraction, sockets will be smoothed and closed with 3-0 silk sutures. Patients will be evaluated on postoperative days 1, 2, 3, and 7 for pain, edema, and trismus. In addition, the control group will receive a dietary supplement containing trypsin, chymotrypsin, and serratiopeptidase (Tripser Forte N30, Incir Pharma, Türkiye), with identical follow-up.
  Interventions: Procedure: Pain Assessment; Procedure: Number of Analgesics Needed; Procedure: Edema Assessment; Procedure: Trismus Assessment

INTERVENTIONS:
Procedure: Pain Assessment — Pain will be assessed using a VAS on the 1st, 2nd, 3rd, and 7th postoperative days. For this purpose, the patient will be shown a 100-mm line with "0" at the left end and "100" at the right end. They will be instructed to mark the point on this line where their pain corresponds. The distance from the marked point to "0" will be measured with a ruler, and the resulting value will be recorded in mm to obtain the VAS score. Changes in these measurements will be recorded.
Procedure: Number of Analgesics Needed — In addition, the number of analgesics required by the patients up to the 7th postoperative day will be recorded.
Procedure: Edema Assessment — To assess edema, the tragus, lateral cauntus, corner of the mouth, and soft tissue pogonion points on the patient's face were marked preoperatively. Preoperatively, on the first, second, third, and seventh postoperative day, measurements will be taken and recorded between the Gonion-corner of the mouth, the Tragus-corner of the mouth, and the Gonion-lateral cauntus points.
Procedure: Trismus Assessment — To assess trismus, the distance between the incisal edges of the upper and lower incisors will be measured and recorded with the mouth maximally open, preoperatively, and on the first, second, third, and seventh postoperative day.

SUMMARY:
Introduction: The aim of this study was to determine the effects of a dietary supplement containing trypsin, chymotrypsin, and serratia peptidase (Tripser Forte N30, Incir Pharma, Turkey) on postoperative healing and to determine the differences between the groups. The aim was to identify differences between the groups regarding postoperative pain, edema, and trismus levels.

Material and Method: Demographic data before surgery will be recorded on the patient follow-up form (Appendix 1). All surgical procedures will be performed under sterile conditions following the administration of local anesthesia (80 mg articaine hydrochloride and 0.02 mg epinephrine, Maxicaine Fort ampoule, Vem Pharmaceuticals, Istanbul, Turkey) with inferior alveolar block anesthesia and buccal mucosa anesthesia. Procedure monitoring will begin after the incision is made and will conclude with suturing. Osteotomy (bone removal) and, if necessary, root dissection will be performed using a surgical handpiece, accompanied by irrigation with sterile saline solution. Following tooth extraction, the socket will be examined, and any sharp bony prominences will be removed. The area will be closed primarily using non-resorbable silk suture material (3/0 surgical silk suture, Doğsan, Turkey). A sterile tampon will be applied to the procedure area, and the patient will be instructed to bite on the tampon for 20 minutes before removing it and replacing it with another material. As a standard postoperative approach, all patients in group 1 received antibiotics (875 mg Amoxicillin+125 mg clavulonic acid, Augmentin-BID film coated tablets, GlaxoSmithKline, Istanbul, Turkey), analgesics (25 mg dexketoprofen, Arveles tb, UFSA Pharmaceutical Industry and Trade Inc. Davutpasa Cad. No.12 (34473) Topkapi/Istanbul) and mouthwash (100 ml solution containing 120 mg (%0.12) chlorhexidine gluconate and 150 mg (%0.15) benzydamine hydrochloride) for use after surgery. Drogsan Pharmaceutical Industry and Trade Inc. Oguzlar neighborhood, 1370.sokak 7/3 Balgat 06520 Cankaya/Ankara). Patients will be instructed to take antibiotics morning and evening for 5 days, use mouthwash for 7 days starting the day after the procedure, and use mouthwash only when deemed necessary. They will be asked to record the amount they use on the provided home assessment form (Appendix 2). Patients in Group 2 will be given a dietary supplement containing trypsin, chymotrypsin, and serratia peptidase (Tripser Forte N30, Incir Pharma, Turkey) in addition to the medications mentioned above. Patient follow-up procedures will be the same.

All patients will be evaluated on the 1st, 2nd, 3rd, and 7th postoperative days, and pain, edema, and trismus will be recorded.

DETAILED DESCRIPTION:
Impacted tooth extractions are the most common clinical procedure in oral and maxillofacial surgery. As with other oral surgical procedures, they are associated with a wide variety of complications, including swelling, pain, limited mouth opening (trismus), bleeding, nerve damage, and delayed healing (1-3). These complications develop following the inflammatory response to the surgical intervention and can be related to factors such as age, gender, systemic condition, position of the impacted tooth, poor oral hygiene, smoking, surgical experience, and duration of the procedure (3). However, the most common complications are pain, swelling, and limited mouth opening. These can lead to a decrease in quality of life, loss of work, and restrictions on social activities (4). To reduce the inflammation that occurs after impacted tooth extraction and to reduce the severity of the aforementioned complications, various medications can be used under the heading of pharmacological methods, or additional non-pharmacological methods such as modified surgical methods, drain placement, low-power laser applications, cold therapy, and physical therapy (5-8). Trypsin, chymotrypsin, and serratia peptidase are proteolytic enzymes and stand out for their various biological functions. The use of these enzymes after surgical interventions such as tooth extraction is being investigated to reduce complications such as postoperative edema, pain, and trismus during the healing process (9).

Proteolytic enzymes such as trypsin, chymotrypsin, and serratia peptidase, when used in conjunction with each other, may contribute to the reduction of postoperative edema, pain, and trismus. Each of these enzymes controls inflammation in different ways, can accelerate the healing process by degrading protein, and promotes faster tissue recovery after surgical trauma (10).

Trypsin is a protease produced by the pancreas and activated in the small intestine. Trypsin contributes to the digestive process by breaking down proteins into peptides and amino acids. Trypsin may help accelerate the healing process, particularly in the body, due to inflammation and tissue damage. This enzyme has effects such as reducing edema, wound healing, and controlling inflammation. It is frequently used after surgical interventions, such as tooth extractions, because it reduces postoperative edema and provides pain relief (11). Studies evaluating the effects of dietary supplements containing trypsin, chymotrypsin, and serratia peptidase after third molar surgery are available in the literature. The primary objective of this study was to clinically evaluate the effects of dietary supplements containing trypsin, chymotrypsin, and serratia peptidase on postoperative edema, pain, and trismus in the postoperative period of mandibular third molar extractions.

ELIGIBILITY:
Inclusion Criteria:

* Having a mandibular third molar with a unilateral or bilateral Class 2, Position A or B impaction according to the Pell and Gregory classification
* Being systemically healthy (ASA Class I)
* Aged between 18 and 45 years (young adult age group)
* Willingness to participate in the study

Exclusion Criteria:

* Age outside the specified range
* Pregnancy
* Currently breastfeeding
* Presence of infection in the third molar region (e.g., acute pericoronitis)
* Presence of cystic or tumoral lesions associated with the impacted third molar
* History of allergic reactions
* Presence of any systemic disease
* Unwillingness to participate in the study
* Poor oral hygiene that may negatively affect healing
* Smoking or alcohol addiction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Wound healing status on postoperative day 7 | Postoperative day 7
  The surgical site will be clinically evaluated for wound healing on day 7 after surgery using a standardized Early Wound Healing Index (EHI), which assesses clinical signs such as redness, swelling, bleeding, and epithelialization. The EHI is scored on a scale from 0 to 5, where 0 indicates very poor healing and 5 indicates excellent healing. Higher scores reflect better healing outcomes. Unit of Measure: Early Wound Healing Index score (0-5)
Change in pain levels after mandibular third molar surgery | From postoperative day 1 to day 7
  Pain levels will be assessed daily for 7 days following mandibular third molar surgery using the Visual Analog Scale (VAS), a 10-centimeter scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity. Patients will complete the VAS form daily, and the average score across the 7-day period will be calculated for each participant. Unit of Measure: Visual Analog Scale score (0-10)
Change in burning sensation levels after mandibular third molar surgery | From postoperative day 1 to day 7
  Burning sensation levels will be assessed daily for 7 days following mandibular third molar surgery using the Visual Analog Scale (VAS), a 10-centimeter scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity. Patients will complete the VAS form daily, and the average score across the 7-day period will be calculated for each participant. Unit of Measure: Visual Analog Scale score (0-10)
Change in facial edema after mandibular third molar surgery | Days 1,2,3 and 7
  Facial edema will be assessed on postoperative days 1, 2, 3, and 7 following mandibular third molar surgery. Swelling will be measured using standardized linear facial measurements obtained with a flexible tape measure between fixed anatomical points (e.g., tragus-oral commissure, tragus-pogonion, and lateral canthus-gonion). The sum of these distances will be recorded at each visit, and the change in facial measurement values over time will be used to evaluate edema. Higher values indicate greater facial swelling.
Change in trismus (maximum mouth opening) after mandibular third molar surgery | Days 1,2,3 and 7
  Trismus will be evaluated on postoperative days 1, 2, 3, and 7 by measuring maximum mouth opening using a calibrated ruler or caliper. Maximum interincisal distance (between the incisal edges of the upper and lower central incisors) will be recorded at each time point. The change in maximum mouth opening over time will be used to assess trismus. Lower interincisal distance values indicate greater trismus.

SECONDARY OUTCOMES:
Number of analgesic tablets consumed postoperatively | From postoperative day 1 to day 7
  Participants will record the number of analgesic tablets taken each day for 7 days after surgery in a home diary. The total number of tablets consumed will be calculated. Unit of Measure: Number of tablets per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient information will be kept confidential.